CLINICAL TRIAL: NCT00466739
Title: European Study of Therapeutic Compliance in Parkinson's Disease
Brief Title: European Compliance Study in Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: South Glasgow University Hospitals NHS Trust (Other)
Responsible Party: Dr D Grosset, Southern General Hospital
Other Study IDs: 05/S0709/95
Record Dates: First submitted 2007-04-26; First posted 2007-04-27 (Estimated); Last update posted 2008-05-23 (Estimated); Status verified 2008-05

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

SUMMARY:
In both symptomatic and asymptomatic disease, only about half of medicines are taken as prescribed1. Relatively little is known about how patients with Parkinson's disease take their medication. One of the challenges in the management of Parkinson's disease is the prevention and treatment of involuntary movements2,3 and wild fluctuations between being mobile and able to function against being slow, stiff and unable to move which recurs as a delayed (several years) effect of taking antiparkinson medication. One theory of why this occurs is that it is due to pulsatile rather than continuous delivery of medication to the brain4. If patients take their medicines erratically and irregularly, this causes more fluctuations in blood and therefore brain drug levels may prime patients for complications in the future. This project will define the extent of irregular medication taking in Parkinson's disease, examine associated clinical and demographic characteristics and examine the ease of adherence to different drug regimes. Knowledge of therapy adherence will help support patients in using their medicines to best effect. In the present document the terms compliance and adherence are used with equal meaning.

DETAILED DESCRIPTION:
This is an observational study of how patients with Parkinson's disease take their medication. Antiparkinson medication will be monitored using electronic pill bottles, MEMS, Aardex®, Switzerland (which contain a microprocessor in the cap that records the time and date of bottle openings). This gives information about the amount of prescribed medication taken (total compliance), the percentage of days when the correct number of doses is taken (daily compliance), and the percentage of doses taken at the correct time interval (timing compliance).

Five countries will be involved, (UK, Germany, Italy, Spain and France). The total number of patients recruited across Europe will be 144. The study size has been calculated based on a single centre study in Glasgow where 2/3 of 120 patients were scheduled to undergo electronic monitoring as part of a different study design. Accordingly data is available which has informed the expected number of patients completing the study (around a 10% drop out rate) and in order to test 6 key variables with potential influence on therapy compliance and using the general statistical guide that between 10 and 20 patients should be studied per variable to be examined, a sample size of around 120 evaluable patients has been calculated.

ELIGIBILITY:
Inclusion Criteria:

* Men or Women between 18 and 80 years.
* Patient has idiopathic Parkinson's Disease according to Brain Bank criteria. - Reference Hughes A J, Daniel S E, Kilford L, Lees A J, Accuracy of Clinical - Diagnosis of Idiopathic Parkinson's disease; A clinical Pathological study of 100 cases, JNNP 1992, 55(3): 181 - 184
* Patient is on stable doses of anti-Parkinson's disease medication, which are not expected to change during the study period.
* Patient is taking levodopa and/or dopamine agonist treatment.
* Patient (assisted by a carer where appropriate) is able to take their medication using the MEMS (electronic monitoring) containers.
* Patients using a dosette box or similar device for their medication are willing to use the MEMS containers for their PD medication
* The investigator judges that the patient's care and symptom control will not be adversely affected by entering the study and using the MEMS device.

Exclusion Criteria:

* Patient is taking anti-Parkinson's disease therapy intermittently or on "as required" basis (such as rescue therapy for off periods). Intermittent Domperidone is allowed.
* Severe co-morbid condition such as severe heart, liver, or kidney disease or cancer diagnosis where the co-morbid condition is of greater health significance than the Parkinson's disease in terms of life expectancy and levels of care required.
* Patient is expected to undergo hospital admission during the study period (such as elective surgery).
* Patient is on non standard drug treatment / combination therapy. This would include e.g. a combination of 2 different oral dopamine agonists, doses of dopamine agonist taken at higher than recommended for routine practice.
* New antiparkinson treatment is being introduced at the time of recruitment or during the one month monitoring period.
* Patient is taking only adjunct therapy (eg. Selegiline, Amantadine, anticholinergic therapy).
* Patient is taking part in a clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Sampling Method: Non-Probability Sample
Enrollment: 144 (Estimated)
Dates: Start 2006-01; Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald Grosset, MD, Principal Investigator — Southern General Hospital, Glasgow, UK
Locations (1):
- Dr D Grosset, Glasgow, United Kingdom